CLINICAL TRIAL: NCT01654237
Title: Factors That Influence the Prevalence of Musculoskeletal Complaints Among Workers in Different Sectors of an Industry
Brief Title: Musculoskeletal Complaints in an Industry
Acronym: FIPMCAWMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 123ERGON; 0344/10 (Registry Identifier: 0344/10)
Record Dates: First submitted 2012-07-27; First posted 2012-07-31 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Musculoskeletal Disorder
Keywords: work; WMSD; prevalence; occupational risks; industry; questionnaires; musculoskeletal pain; lifestyle
MeSH Terms: conditions — Musculoskeletal Diseases; Musculoskeletal Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Muskind (No Intervention): three questionnaires to be completed by the subjects
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — 185 industry workers divided in three sectors (factory, office and logistics) were assessed using the Nordic Musculoskeletal Questionnaire and lifestyle and work-related conditions questionnaires.

SUMMARY:
The hypothesis of this study is that there will be a variety of factors influencing the musculoskeletal complaints among workers of different sectors.

Work-related musculoskeletal disorders (WMSDs) account for more than 30% of occupational diseases in the world. In order to organize the strategic actions that will be developed for the prevention of MSDs, it is essential to analyze in advance the peculiar situations of the different sectors of a workplace. The objectives of this study were to determine the prevalence of musculoskeletal complaints among workers in a medium-sized industry by comparing its sectors and to investigate the influence of occupational and non-occupational factors in the increase of complaints.

DETAILED DESCRIPTION:
The Nordic questionnaire was used to asses musculoskeletal symptoms as well as questionnaires about lifestyle and work-related conditions in 185 workers divided into three sectors of an industry (factory - microelectronics, office and logistics)

ELIGIBILITY:
Inclusion Criteria:

* work in the industry

Exclusion Criteria:

* work less than a month in the industry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
musculoskeletal complaints | one month
  musculoskeletal complaints in different parts of the body

CONTACTS AND LOCATIONS:
Overall Officials: Denise Harari, post grad, Principal Investigator — Faculty of Medicine. University of Sao Paulo; Raquel A Casarotto, doctor, Study Director — Faculty of Medicine. University of Sao Paulo
Locations (1):
- Faculty of Medicine. University of Sao Paulo, São Paulo, Sao Paulo/SP, Brazil